CLINICAL TRIAL: NCT05452200
Title: Pilot Study on Lung Cancer Screening Implementation Among Employees at Lyon Hospital
Brief Title: Lung Cancer Screening Implementation Among Employees at Lyon Hospital
Acronym: ILYAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0466
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
Keywords: lung cancer; screening; tobacco cessation; COPD
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Cessation; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lyon hospital employees with high risk of lung cancer. (Experimental): Lyon Hospital employees meeting criteria for high risk of lung cancer according French recommendation criteria.
  Interventions: Behavioral: Solicitation for lung cancer screening; Other: added exams to the usual lung cancer screening

INTERVENTIONS:
Behavioral: Solicitation for lung cancer screening — 3 levels of solicitation will be cumulated. First : a Simple collective solicitation of all staff via internal media 4 months later : Personalized indirect solicitation of at-risk groups with information posted in identified areas 4 months later : Personalized direct solicitation of at-risk groups
Other: added exams to the usual lung cancer screening — * spirometry examination
  * Questionnaires
  * Blood samples and breath samples to find biomarkers

SUMMARY:
Several randomized studies have demonstrated the efficiency of lung cancer screening (LCS) on mortality rates. However, screening efficiency is related to the targeted population and the participation rate.

In France, the participation rate for breast and colon cancer screening programs is respectively 50% and 32%, which is low. Then, it appears very important to determine which factors are influencing the willingness to participate to these programs. Indeed, it will allow a better communication and we will be able to perform screening campaigns adapted to the eligible population.

The Lyon Hospital is the second university hospital in France. It is composed of 14 buildings and employed 23 000 persons. More than 160 occupations are represented. So, hospital employees look relevant to be studied for LCS program.

ILYAD was divided in 2 parts. The first one was completed in 2020 and goal to evaluate the number of eligible individuals among the hospital employees. About 800 persons would be eligible for LCS.

This second part of the study will evaluate the participation rate and the feasibility of the LCS program. The study will target the 800 individuals that were identified previously.

ELIGIBILITY:
* Inclusion Criteria :

  * Participant have to meet the criteria below:

Lyon hospital employee at the day of inclusion:

* valid hospital employee number,
* Or retired employee for less than a year before the inclusion

AND meeting eligibility criteria as follow :

* Aged from 50 to 75 yo,
* AND smoke or have smoked ≥ 10 cigarettes/day during ≥ 30 years OR ≥ 15 cigarettes/day for at least 25 years;
* AND active smoker or smoking cessation for ≤ 15 years ;

  * Volunteer to start a program of smoking cessation if active smoker;
  * Consent form signed ;
  * Cover by health insurance.

    * Exclusion Criteria :

Participant have to NOT meet the criteria below :

* Individual not working at Lyon hospital;
* Individual not payed by the Lyon Hospital but working at it;
* Individuals not willing to participate;
* Individual working at René Sabran Hospital;
* Individual meeting one of this non eligibility for LCS criteria defined by the French recommendation:

  * Not able to climb 2 floors of stairs ;
  * Weight ≥ 140Kg
  * Underwent a chest CT scan less than 1 year ago (except screening scanner);
  * History of lung cancer of less than 5 years or under treatment ; history of any cancer under monitoring by chest scanner ;
  * Comorbidity contraindicating therapeutic options or any kind of invasive interventions ;
  * Ongoing or recent respiratory symptoms that might lead to lung cancer diagnosis (hemoptysia, weight loss, recurrent respiratory infection).
* Individual who is pregnant or breast feeding;
* Individual whose mental health is not good enough to participate;
* Individual in jail or under justice evaluation.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-09-12 (Estimated); Study Completion 2024-09-12 (Estimated)

PRIMARY OUTCOMES:
Participation rate at baseline | At the baseline visit
  Ratio between the number of participants who underwent a CT scan at baseline and the estimated number of eligible employees

SECONDARY OUTCOMES:
Participation rate according to the 3 communication levels. | At 4 month = level 1 ; At 8 month = level 2 ; At 12 month = level 3
  Ratio between the number of participants who underwent the baseline CT scan at level 1, 2 and 3 and the estimated number of eligible employees
Identification of predictive factors for participation decision | At baseline and At 1Year follow-up
  Using the cox model to identify sociodemographic factors that could be associated with the participation rates for both round of CT scan.
Evaluation of feasibility of the LCS program by measuring the proportion of individuals having undergo all the required exams and evaluations according to the results of the CT scan, conformity of the scan interpretation, and adverse event monitoring. | At baseline and At 1Year follow-up
  Ratio between individuals who completed baseline and year 1 CT scan and the number of participants. And, the ratio of individuals who beneficiated conform care according to French recommendations.
Evaluation of screening efficiency according to the proportion of lung cancer, ILD, COPD diagnosed and the percentage of smoking cessation among the active smokers. | At baseline and At 1Year follow-up
  Ratio of lung cancer diagnosed Ration of ILD diagnosed Ratio of COPD diagnosed Ratio of smoking cessation
Evaluate the participation rate at 1 year and identify the factors that trigger it. | At 1Year follow-up
  Ratio between the number of participants who underwent the Year 1 CT scan and the number of participants.
Identification of efficient biomarker for LC screening | At baseline
  Perform blood analysis to identify specific biomarkers and compare their sensibility, and predictive value with or without association with the CT scan.
Evaluation of the efficiency of VOC for LC screening | At baseline
  Perform air breath analysis to identify specific chemical species, compare their sensibility, and predictive value associated, and not with the CT scan.
Evaluate the follow up to the french guidelines | Follow up after the 1 year visit
  Ratio between the participant at the cohort and who have done the scanner 2 years post Year1 one, and the participant at the cohort.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital L. Pradel, Bron
  - Hôpital de la Croix Rousse - Department of Pneumology, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No